CLINICAL TRIAL: NCT02444104
Title: Validation of Non-invasive Blood Pressure and Cardiac-output Measurement by Using Applanation Tonometry in Cardiological Patients
Brief Title: Non-invasive Blood Pressure and Cardiac Output Measurement by Using Applanation Tonometry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: TNSYS2015
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Atrial Fibrillation; Left Ventricular Failure; Left Ventricular Impaired Function; Aortic Valve Stenosis
Keywords: Left Ventricular Assist Device
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients with atrial fibrillation: It is Primarily a comparison of methods , non-invasive measured blood pressure versus invasively measured blood pressure and non-invasively measurement of cardiac output versus invasive cardiac output measurement in patients with atrial fibrillation.
- Patients with highly reduced LV function: It is Primarily a comparison of methods , non-invasive measured blood pressure versus invasively measured blood pressure and non-invasively measurement of cardiac output versus invasive cardiac output measurement in patients with a highly reduced left ventricular function (LV function)
- Patients with aortic stenosis: It is Primarily a comparison of methods , non-invasive measured blood pressure versus invasively measured blood pressure and non-invasively measurement of cardiac output versus invasive cardiac output measurement in patients with severe aortic stenosis
- Patients with LVAD: It is Primarily a comparison of methods , non-invasive measured blood pressure versus invasively measured blood pressure and non-invasively measurement of cardiac output versus invasive cardiac output measurement in patients with left ventricular assist-device (LVAD)

SUMMARY:
To evaluate and to validate accuracy, precision and trending ability of blood pressure and cardiac output measurement by applanation tonometry in cardiological patients having:

* atrial fibrillation
* severe impaired leftventricular function
* severe aortic valve stenosis
* patients having left ventricular assist device

Experimental measurement: continuous blood pressure measurement and cardiac output measurement is performed by the T-Line 200 pro device (Tensys Medical Inc., San Diego, USA) Control measurement: gold-standard continuous blood pressure measurement is performed by invasive blood pressure measurement by arterial cannulation and cardiac output reference is assessed by transcardiopulmonary thermodilution

DETAILED DESCRIPTION:
Increasing complexity of medical interventions and critical care treatment in an elderly getting population requires precise and accurate hemodynamic monitoring.(1) However, advanced invasive hemodynamic monitoring is often combined with complications by arterial or central venous catheterization. Complications such as vessel harming, infection, cardiac arrhythmias and nervous lesions are likely to occur.(2-4) Therefore, in the past various techniques of minimal- or non-invasive hemodynamic monitoring devices have been evaluated.(5, 6) One of the very promising technique is continuous non-invasive blood pressure monitoring by applanation tonometry. Published data revealed efficacy of this technique. (7) However, ability of this technique remains unclear in patients suffering from cardiological pathologies leading to changing stroke volumes as in arterial fibrillation, to highly reduces stroke volume as in severe impaired left-ventricular function or in severe aortic valve stenosis. Further, ability of applanation tonometry in patients without having pulsatile blood flow such as in patients with left-ventricular assist device remains unclear. Therefore, validation of this technique should be performed in the presented study.

Further development of applanation tonometry including pulse contour analysis now enables assessment of cardiac output. However, till now there is limited data assessing validation cardiac output measurement by this method. Cardiac output validation should also be performed in the planed clinical study.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation
* severe impaired leftventricular function
* severe aortic stenosis
* LVAD Patients

Exclusion Criteria:

* Age <18 years
* pregnancy
* patients having blood pressure difference of more than 10 mmHg on both arms (measurement by "Riva-Rocci" before study enrolment)
* pre-existing on arterial vessels of the arms
* patients who are not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enable for study enrollement need to suffer from one of the four cardiological pathologies:
  1. atrial fibrillation,
  2. severe impaired leftventricular function,
  3. severe aortic valve stenosis
  4. patients having left ventricular assist device
  All patients have to be clinically monitored by invasive blood pressure assessment and transcardiopulmonary thermodilution.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy and precision of blood pressure and cardiac output by applanation tonometry | 30 minutes

SECONDARY OUTCOMES:
Trending ability of blood pressure monitoring by applanation tonometry | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Reuter, Study Director — University Hamburg
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Saugel B, Reuter DA. Are we ready for the age of non-invasive haemodynamic monitoring? Br J Anaesth. 2014 Sep;113(3):340-3. doi: 10.1093/bja/aeu145. Epub 2014 May 31. No abstract available. PMID 24880826
- [Background] Mandel MA, Dauchot PJ. Radial artery cannulation in 1,000 patients: precautions and complications. J Hand Surg Am. 1977 Nov;2(6):482-5. doi: 10.1016/s0363-5023(77)80030-0. PMID 925335
- [Background] Russell JA, Joel M, Hudson RJ, Mangano DT, Schlobohm RM. Prospective evaluation of radial and femoral artery catheterization sites in critically ill adults. Crit Care Med. 1983 Dec;11(12):936-9. doi: 10.1097/00003246-198312000-00007. PMID 6641252
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Reuter DA, Huang C, Edrich T, Shernan SK, Eltzschig HK. Cardiac output monitoring using indicator-dilution techniques: basics, limits, and perspectives. Anesth Analg. 2010 Mar 1;110(3):799-811. doi: 10.1213/ANE.0b013e3181cc885a. PMID 20185659
- [Background] Saugel B, Trepte CJ, Heckel K, Wagner JY, Reuter DA. Hemodynamic management of septic shock: is it time for "individualized goal-directed hemodynamic therapy" and for specifically targeting the microcirculation? Shock. 2015 Jun;43(6):522-9. doi: 10.1097/SHK.0000000000000345. PMID 25643016
- [Background] Saugel B, Meidert AS, Hapfelmeier A, Eyer F, Schmid RM, Huber W. Non-invasive continuous arterial pressure measurement based on radial artery tonometry in the intensive care unit: a method comparison study using the T-Line TL-200pro device. Br J Anaesth. 2013 Aug;111(2):185-90. doi: 10.1093/bja/aet025. Epub 2013 Mar 13. PMID 23491946